CLINICAL TRIAL: NCT01611662
Title: Phase II Trial of Neoadjuvant Dose Dense Gemcitabine and Cisplatin In Muscle Invasive Bladder Cancer
Brief Title: Gemcitabine Hydrochloride and Cisplatin Before Surgery in Treating Patients With Muscle Invasive Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme Toxicity
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERP-GU-052; NCI-2012-00906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB#12-015 (Other: Fox Chase Cancer Center); ERP-GU-052 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Distal Urethral Cancer; Proximal Urethral Cancer; Squamous Cell Carcinoma of the Bladder; Stage II Bladder Cancer; Stage III Bladder Cancer; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine hydrochloride, cisplatin, surgery) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on day 1 and cisplatin IV on day 1 or divided over days 1 and 2. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-8 weeks after chemotherapy, patients undergo radical cystectomy.
  Interventions: Drug: gemcitabine hydrochloride; Drug: cisplatin; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Procedure: therapeutic conventional surgery — Undergo radical cystectomy
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this research study is to find out what effects, good and/or bad, dose-dense (every 14 days) chemotherapy with gemcitabine (gemcitabine hydrochloride) and cisplatin given before surgery have on patients and their muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of complete response (pT0) at cystectomy following preoperative dose dense gemcitabine and cisplatin (DD GC) in patients with muscle invasive urothelial carcinoma of the bladder.

SECONDARY OBJECTIVES:

I. To assess the toxicity profile of DD GC when given in the neoadjuvant setting: To define the number of patients who complete all three cycles of treatment without dose reduction, and to describe the incidence of toxicity.

II. To assess the 5 year overall and relapse free survival in patients who receive neoadjuvant DD GC.

TERTIARY OBJECTIVES:

I. To evaluate tissue specimens from patients to assess for molecular markers that correlate with clinical outcome.

OUTLINE:

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on day 1 and cisplatin IV on day 1 or divided over days 1 and 2. Treatment repeats every 14 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-8 weeks after chemotherapy, patients undergo radical cystectomy.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed urothelial carcinoma of the bladder or urethra; patients with urothelial carcinoma of the prostatic urethra only may be included at primary investigator (PI) discretion; T-stage must be T2 to T4a; patients with radiographic N0 disease or N1 disease are eligible for the study; patients must not have radiographic evidence of metastatic disease; mixed histologies which are predominantly urothelial, such as with squamous or micropapillary differentiation, are allowed so long as there is no component of small cell histology; histology must be confirmed by a pathologist at an institution involved in this study
* Patients must be candidates for radical cystectomy with the goal of cure
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN
* Patients must have adequate renal function defined as creatinine clearance >= 50 mL/min; for eligibility, creatinine clearance may be either calculated using the Cockcroft-Gault formula or measured with 24 hour urine collection; note that 24 hour urine collection is required at baseline, but does not have to be used for eligibility if calculated clearance by Cockcroft-Gault is preferred; nephrostomy or ureteral stent placement in order to achieve adequate creatinine clearance is allowed
* Women of child-bearing potential (WOCBP) and men with a female partner who is a WOCBP must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) starting prior to beginning treatment and continuing until at least 3 months after last dose of chemotherapy and surgery; should a woman become pregnant or suspect she is pregnant while participating in this study or if a female partner of a man participating in this study becomes pregnant, the treating physician must be notified immediately; WOCBP must have a negative serum or urine pregnancy test within 7 days prior to initiating study treatment
* No other active malignancy
* Ability to understand and the willingness to sign written informed consent and Health Insurance Portability and Accountability Act (HIPAA) documents

Exclusion Criteria:

* Patients who have had intravesicular therapy within 4 weeks of study entry, or those who have not recovered from adverse effects of such agents administered more than 4 weeks earlier
* Patients may not be receiving any investigational agents within 4 weeks of study entry
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or cisplatin or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have undergone prior radiation to greater than or equal to 25% of the bone marrow within the past year are excluded
* Patients who have received any previous systemic chemotherapy or radiation therapy for urothelial carcinoma within 1 year of study entry are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2013-07-12 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Plimack, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Thomas Jefferson University, Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Satyal U, Valentine H, Liu D, Slifker M, Lallas CD, Trabulsi EJ, Bukavina L, Szeto L, Hoffman-Censits JH, Mouw KW, Faltas BM, Grivas P, Ibragimova I, Porten SP, Van Allen EM, Geynisman DM, Parker DC, O'Neill JP, Drevik J, Christianson SS, Ginzburg S, Correa AF, Uzzo RG, Ross EA, Zibelman MR, Ghatalia P, Plimack ER, Kutikov A, Abbosh PH. Urine Biopsy as Dynamic Biomarker to Enhance Clinical Staging of Bladder Cancer in Radical Cystectomy Candidates. JCO Precis Oncol. 2024 Jun;8:e2300362. doi: 10.1200/PO.23.00362. PMID 38865671

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery)
Started | 32
Completed | 31
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: The tumor in patients was graded by TNM staging where T refers to the stage of primary tumor, n refers to the regional lymph nodes, M refers to distant metastasis. T0 - no evidence of primary tumor; N0- no regional lymph nodes; M0-no distant metastasis
Arm/Group | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21
Baseline clinical stage [Count of Participants; unit: Participants]
  T2N0M0 | 11
  T3N0M0 | 15
  T4aN0Mo/TxN1M0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response Rate Following Chemotherapy Before Surgery
Description: Pathological response rate following neoadjuvant chemotherapy was assessed by TNM staging at the time of radical cystectomy
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery)
Number analyzed (Participants) | 31
percentage of participants | 32 [16 to 48]

ADVERSE EVENTS:
Arm/Group | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery)
Serious Adverse Events (participants affected / at risk) | 16/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery) (N=31)
Chest pain (Cardiac disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 2
Acute Kidney Injury (Renal and urinary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Acute Renal Insufficiency (Blood and lymphatic system disorders) | 1
Coronary Artey Disease (Cardiac disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
hypotension (Vascular disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
infected lymphocele (Infections and infestations) | 1
Fever (General disorders) | 3
Nausea (Gastrointestinal disorders) | 1
bacteremia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
hyperkalemia (Metabolism and nutrition disorders) | 2
hypernatremia (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
vomiting (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Gout (Musculoskeletal and connective tissue disorders) | 1
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
cerebral Infarction (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Gemcitabine Hydrochloride, Cisplatin, Surgery) (N=31)
Anemia (Blood and lymphatic system disorders) | 29
Atrial Fibrilation (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 1
Sinus Brachycardia (Cardiac disorders) | 1
Sinus Trachycardia (Cardiac disorders) | 4
Cardiac Faliure (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Hearing Impaired (Ear and labyrinth disorders) | 1
Blurred Vision (Eye disorders) | 1
Tinnitus (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 1
GERD (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 24
vomiting (Gastrointestinal disorders) | 5
chills (General disorders) | 5
Edema (General disorders) | 6
fatigue (General disorders) | 30
fever (General disorders) | 5
flu-like symptoms (General disorders) | 2
infusion related reaction (General disorders) | 2
pelvic pain (Reproductive system and breast disorders) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
AST/SGOT (Investigations) | 3
Injection site reaction (General disorders) | 3
ALT/SGPT (Investigations) | 4
Alkaline Phosphatase increased (Investigations) | 15
blood bilirubin increased (Investigations) | 1
creatinine increased (Investigations) | 15
White blood cells decreased (Investigations) | 4
ANC decreased (Investigations) | 4
Platelet count decreased (Investigations) | 9
lymphocyte count decreased (Investigations) | 13
cardiac troponin increased (Investigations) | 3
Weight loss (Investigations) | 2
Dehydration (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 12
Hypokalemia (Metabolism and nutrition disorders) | 14
Hypernatremia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 24
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesium (Metabolism and nutrition disorders) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 12
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 10
Acute kidney injury (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Infection (Infections and infestations) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 3
extravasation (General disorders) | 1
lymphocele (Vascular disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Phlebitis (Infections and infestations) | 2
intra-abdominal infection (Infections and infestations) | 1
urinary retention (Renal and urinary disorders) | 1
Glaucoma (Eye disorders) | 1
Infusion site extravasation (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No